CLINICAL TRIAL: NCT02155777
Title: Mechanisms of Prevention of Ovarian Cancer by Oral Contraceptives
Brief Title: Why do Oral Contraceptives Prevent Ovarian Cancer?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Celeste Pearce, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OC Prevention; 1R21CA178571-01 (NIH)
Record Dates: First submitted 2014-05-15; First posted 2014-06-04 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Ovarian Cancer Risk; Risk-reducing Surgery; Fallopian Tube Fimbriae; Ovarian Cortical Inclusion Cysts
Keywords: BRCA1; BRCA2; Risk-reducing surgery; Oral Contraceptives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention): No intervention.
- OrthoNovum 1/35 (Active Comparator): OrthoNovum 1/35
  Interventions: Drug: OrthoNovum 1/35

INTERVENTIONS:
Drug: OrthoNovum 1/35
  Arms: OrthoNovum 1/35

SUMMARY:
Use of oral contraceptives (OCs) reduces a woman's risk of ovarian cancer very significantly and the protective effect continues for at least 25 years after use of OCs is stopped; the mechanisms of how this occurs are not understood. We are proposing here to directly study the effect of OCs on the fallopian tube and inclusion cysts within the ovary - sites from which most ovarian cancers are thought to arise - in order to better understand the mechanistic basis for OC protection against ovarian cancer. We think the protection results from reduced cell proliferation. It will lay the foundation for further studies to ensure that the protection against ovarian cancer afforded by 'traditional' OCs is not lost with alterations in OC formulation, and, if possible, to guide development of OC formations to improve further on the protection afforded by OCs.

DETAILED DESCRIPTION:
Five-year survival for invasive epithelial ovarian cancer (ovarian cancer) is less than 50% because most women are diagnosed at an advanced stage. However, there is an effective chemoprevention strategy. Meta-analysis of epidemiological studies shows an approximately 40% reduction in risk of ovarian cancer with 5 years of oral contraceptive (OC) use. The protective effect increases significantly with duration of OC use and continues for at least 25 years after use of OCs is stopped. The mechanism(s) underlying this protective effect are not understood. One hypothesis is that protection is achieved by blocking ovulation, but growing evidence suggests that it may be related to promoting a favorable progestagenic environment. OC use would protect if the hormonal exposure while on OCs was less stimulatory to the possibly different types of cells of origin of ovarian cancer than the hormonal exposure in normal ovulatory cycles. Exposure to progestins is higher while on OCs than in normal cycling and this could explain the protective effect. We propose that a major source of the protection from OC use is due to their significantly reducing cell proliferation in the fallopian tube fimbriae (FTF) and in ovarian cortical inclusion cysts (CICs), two likely cells of origin for ovarian cancer. Proliferating cell populations are more susceptible to carcinogenic effects with the rise in cancer risk with cell proliferation being secondary to increased chances of mutation and progression. FTF proliferation has been reported to be almost confined to the follicular phase of the menstrual cycle with virtually no proliferation within a few days after ovulation and our preliminary data show the same pattern - OCs could thus protect against ovarian cancers arising in the FTF by mimicking the luteal phase of the cycle when progesterone exposure is high. Whether such changes occur in CICs is not known. Cell proliferation within different types of CICs during the menstrual cycle has not been studied. The effect of OCs on proliferation within the FTF and CICs has also not been studied. We are proposing to determine the effect of a 'traditional' high progestin dose OC on cell proliferation in the FTF and CICs in women undergoing a risk-reducing bilateral salpingo-oophorectomy (RR-BSO), and to compare these proliferation rates to the rates during the normal menstrual cycle of women also undergoing an RR-BSO. The results of this study will provide crucial information regarding the relationship between OC use and protection against ovarian cancer. It will lay the foundation for further studies examining the effects of lower progestin dose OCs and OCs with newer progestin formulations. Our long-term goal in studying the mechanism of OC protection is to determine whether it is likely that the protection against ovarian cancer afforded by OCs will be lost with alterations in OC formulation in terms of dose or type of progestin used, and, if possible, to guide development of OC formations to improve further on the protection afforded by OCs.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* 30 and 45 years of age
* Scheduled to undergo a laproscopically conducted RR-BSO, risk reducing salpingectomy, salpingectomy for sterilization, or salpingectomy with hysterectomy for non-cancer related conditions
* Have at least one ovary

Exclusion Criteria:

* Past hysterectomy
* Past diagnosis of ovarian cancer
* Use of Tamoxifen, Raloxifene or hormone replacement therapy in the past 3 months
* Use of Chemotherapy in the last 6 months

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Differences in cell proliferation as measured by Ki67 immunohistochemical analysis in the fallopian tube fimbriae of women on the OC arm compared to women on the no treatment arm. | Cell proliferation (Ki67) will be measured in the specimen that is removed as part of the patients surgery (the surgery is not a study procedure).

SECONDARY OUTCOMES:
Cell proliferation as measured by Ki67 immunohistochemical analysis in ovarian cortical inclusion cysts of women on the OC arm compared to women on the no treatment arm. | Cell proliferation (Ki67) will be measured in the tissue removed as part of the surgery (the surgery is not a study procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste L Pearce, PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (2):
  - USC Keck School of Medicine, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
- UBC BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No